CLINICAL TRIAL: NCT02870699
Title: Study of the Effectiveness of the Film-forming Solution Evonail® Versus Placebo in the Prevention of Nail Damage Induced by Docetaxel in Patients With Breast Cancer.
Brief Title: Efficacy of Evonail® Solution in the Prevention of Nail Damage Induced by Docetaxel in Patients With Breast Cancer.
Acronym: EVONAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-A00981-40
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2018-08

CONDITIONS: Breast Carcinoma
Keywords: chemotherapy neoadjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): * Evonail film forming solution : 1 daily application on the left hand
  * Placebo excipient : 1 daily application on the right hand
  Interventions: Device: Evonail; Device: Placebo excipient
- ARM B (Active Comparator): * Evonail film forming solution : 1 daily application on the right hand
  * Placebo excipient : 1 daily application on the left hand
  Interventions: Device: Evonail; Device: Placebo excipient

INTERVENTIONS:
Device: Evonail — film-forming solution containing water Evaux naturally rich in lithium, strontium and manganese with UV filter
Device: Placebo excipient — film forming excipient solution

SUMMARY:
Docetaxel is widely used in oncology for the treatment of many solid tumors. The side effects of docetaxel are many and sometimes serious. The primary toxicity of docetaxel is neutropenia. Skin and nail manifestations, frequency, the second category of adverse events after haematological adverse events.

Use of the product Evonail® was demonstrated in a patient treated by doxetaxel and having nail damage.

The purpose of this study is to confirm the effectiveness of the film-forming solution Evonail® versus a placebo on the prevention of nail damage in women with breast cancer and treated by adjuvant docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with breast carcinoma
* Patients treated with adjuvant chemotherapy (FEC + 3 docetaxel +/- Herceptin®)
* Patients who have never been treated with taxanes
* Patients with no nail damage before starting the study
* ECOG performance < 2
* Ability to provide written informed consent

Exclusion Criteria:

* Patient allergic to any of the treatment components
* Use of film-forming solution, solvents or any other products applied to the fingernails (artificial nails ...) in three weeks before the first of docetaxel treatment
* Risk of exposure to aggressive factors nail during the study
* Using refrigerants gloves during chemotherapy treatments
* Onychophagia
* Presence of nail disease or a history of nail pathology (infectious and other)
* Pregnant or breast feeding females
* Patients whose condition is not compatible with the follow-up study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of the film-forming solution Evonail® versus placebo on nail damage | up to 9 weeks
  Efficacy will be evaluated by the oncologist according to NCI-CTC

SECONDARY OUTCOMES:
Different types of nail damage observed in each group after chemotherapy docetaxel | up to 9 weeks
  Nail damage will be evaluated by the dermatologist based on photography according to NCI-CTC
Patient compliance for the film-forming solution Evonail® | up to 9 weeks
  Patient compliance will be evaluated using a questionnaire
Patient satisfaction regarding the use of the film-forming solution Evonail® | up to 9 weeks
  Patient satisfaction will be evaluated using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: UWER Lionel, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No